CLINICAL TRIAL: NCT01923298
Title: A Single-arm Phase II Trial to Evaluate Serum Estradiol Levels in Patients With Breast Cancer Treated With Vaginal Estrogen, Estring
Brief Title: Estradiol Levels in Patients Treated With Estring
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-0477-04; EString (Other: The University of Arizona Cancer Center)
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Results first posted 2022-02-04 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Estrogen Levels Among Breast Cancer Patients
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Estradiol (Experimental): ESTRING® (estradiol vaginal ring) is a slightly opaque ring with a whitish core containing a drug reservoir of 2 mg estradiol. Estradiol, silicone polymers and barium sulfate are combined to form the ring. When placed in the vagina, ESTRING releases estradiol, approximately 7.5 mcg per 24 hours, in a consistent stable manner over 90 days.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol
  Other Names: ESTRING®

SUMMARY:
Estrogen receptor positive breast cancer is the most common type of breast cancer and anti-estrogen therapy has been shown to be very effective in preventing recurrence. Side effects of anti-estrogens are due to estrogen deprivation and include hot flashes, mood changes and vaginal dryness/pain. Vaginal symptoms including pain, dryness, itching, bleeding after intercourse and frequent urinary tract infections have been reported to cause significant morbidity in postmenopausal women and higher in breast cancer survivors on anti-estrogen therapy. Treatment options include vaginal lubricants, Replens etc but unfortunately many women continue to have persistent symptoms. Local estrogen has been shown to be effective in post menopausal women (Estring or Vagifem) for their vaginal symptoms. There is a concern of using this in women with breast cancer given it may increase their blood estrogen levels. Studies done so far show have shown controversial results but majority of them report that blood estrogen levels do not change significantly. The major drawback of the studies was the sample size and inadequate accrual. The most recent trial reported showed no significant change in blood estrogen levels in women with breast cancer treated with aromatase inhibitors (anti-estrogen therapy) and were on vagifem for their vaginal symptoms. The authors reported results in 26 patients and reported no significant change in blood estrogen level. We propose to study the change in blood estrogen level when postmenopausal women with breast cancer who are currently on aromatase inhibitors are treated with Estring for their vaginal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III estrogen receptor positive breast cancer (positive for estrogen receptor (ER)) with positivity defined as immunohistochemical staining in ≥ 10% of cells) on adjuvant hormonal therapy with aromatase inhibitors (anastrozole, letrozole or exemestane)
* Adults over 18 years of age with a life expectancy of at least 3 months
* Attained menopause as defined by World Health Organization Criteria (defined as permanent cessation of menstruation resulting from the loss of ovarian follicular activity. This is recognized to occur after 12 consecutive months of amenorrhea, for which there is no other obvious pathological or physiological cause.)
* Persistent genitourinary symptoms causing discomfort for more than 2 weeks prior to the visit with the physician.
* Tried at least 1 prior pharmacological/ non-pharmacological treatment for their genitourinary symptoms
* Be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to any study specific procedures
* Be willing and able to comply with the treatment plan, scheduled clinic visits, laboratory tests and other study procedures

Exclusion Criteria:

* Patients with metastatic breast cancer
* Have a concurrent active non-breast malignancy except for non-melanoma skin cancer
* Patients with vaginal stenosis
* Patients unable to apply Estring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08-09 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Result] Streff A, Chu-Pilli M, Stopeck A, Chalasani P. Changes in serum estradiol levels with Estring in postmenopausal women with breast cancer treated with aromatase inhibitors. Support Care Cancer. 2021 Jan;29(1):187-191. doi: 10.1007/s00520-020-05466-1. Epub 2020 Apr 23. PMID 32328775

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Estradiol
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Estradiol
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 55 [41 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum Estradiol
Description: To measure changes in serum estradiol level compared to their baseline in patients with breast cancer when treated with vaginal estrogen preparation, Estring
Time Frame: Baseline, 16 weeks
Population: Eligible patients were 18 years or older, diagnosed with HR-positive breast cancer defined as > 1% of tumor cells expressing estrogen or progesterone receptors, attained menopause as defined by the World Health Organization, and on adjuvant hormonal therapy with an aromatase inhibitor- anastrozole, letrozole, or exemestane. Patients with metastatic disease were excluded.
Measure: Median (Full Range); unit: pg/mL
Groups:
- Estring Group: ESTRING® (estradiol vaginal ring) is a slightly opaque ring with a whitish core containing a drug reservoir of 2 mg estradiol. Estradiol, silicone polymers and barium sulfate are combined to form the ring. When placed in the vagina, ESTRING releases estradiol, approximately 7.5 mcg per 24 hours, in a consistent stable manner over 90 days.
Arm/Group | Estring Group
Number analyzed (Participants) | 14
pg/mL | 3.9 [1.1 to 8.9]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed through study completion.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed through study completion.
Arm/Group | Estradiol
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT01923298/Prot_SAP_000.pdf